CLINICAL TRIAL: NCT01167842
Title: Analysis of Inherited Cancers
Brief Title: Analysis of Tumors From Patients With Inherited Cancers Having Had Two Surgeries (Primary + Recurrent, or 2 Separate Types of Cancer)
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Elizabeth Swisher, Associate Professor, Obstetrics & Gynecology, University of Washington
Other Study IDs: 7016; P50CA083636 (NIH)
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — We will collect blood as a source for DNA from lymphocytes as well as tumor blocks as a source for tumor DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will analyze tumor tissue from patients with known genetic mutations (BRCA1, BRCA2, CHK2, etc) who have tumor tissue available from two surgeries, either primary/recurrent, or two different anatomical sites.

DETAILED DESCRIPTION:
This study will recruit individuals with known BRCA1 and BRCA2 mutations or mutations in similar cancer causing genes such as CHK2 or PALB2 who have had a cancer removed by surgery or biopsied two or more times with available pathological blocks. We wish to enroll individuals who have had more than one surgery or biopsy for cancer allowing us to obtain tumor blocks from more than one time point. Such patients would include those with one cancer which has recurred or more than one separate cancer. We will conduct a brief interview with the subject to obtain personal information about medical and treatment history. In addition, we will collect clinical information from their treating physician(s) to correlate molecular findings with clinical responses to treatment and survival and recurrence data. We will collect background clinical information and family history information and a copy of the genetic test results documenting their cancer causing mutation. We will recruit only patients with known BRCA1 or BRCA2 mutations or known mutations in other cancer causing genes such as CHK2 or PALB2 and will not perform genetic testing on non-tumor tissue for any new information on genetic susceptibility in patient samples. Enrolled subjects will donate a blood sample that will be obtained locally and shipped to the research laboratory, and this cost will be entirely covered by the research group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 or older
* documented mutation in BRCA1, BRCA2 or other known cancer causing gene
* one or more cancer with available stored tissue blocks or slides
* willing to donate 16cc of blood
* able to understand English and provide informed consent

Exclusion Criteria:

* unable or unwilling to provide informed consent
* patient does not have tissue blocks available
* minor, under age 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, Cancer center, University medical center
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Analysis of Inherited Cancers | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Swisher, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States